CLINICAL TRIAL: NCT03954847
Title: Clinical Significance of Computer Aided Image Analysis in Treatment Response Evaluation of Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: WuhanUH-V1.2
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Image; Treatment response; Prognosis; Radiomic; Deep learning
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung cancer patients: Lung cancer patients with PET/CT or CT examination before any cancer-specific treatment

SUMMARY:
The investigators will evaluate the utility of computer aided image analysis in lung cancer with the aim of predicting treatment response and prognosis.

DETAILED DESCRIPTION:
Tumor biological behavior is the fundamental cause of heterogeneous prognosis. The features found on medical images are also reflections of the tumor biological behavior. However, the limitations in spatial and intensity resolution of the naked eye are two inevitable shortcomings of image interpretation by naked eyes, resulting in subjective and limited analyses of images. Computer aided image analyses such as radiomic analysis and machine learning methods are emerging as promising image interpretation methods. The natural advantage of the unlimited spatial and intensity resolution of computers can overcome the shortcomings of visual inspection with the naked eye. Moreover, the massive computing power of computer is also far greater than that of humans. This study will focus on the application of computer aided analysis in predicting treatment response and prognosis in lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >= 18 years old
2. Pathological diagnosis of NSCLC between 2012 and 2019;
3. PET/CT or CT examination before any cancer-specific treatment;

Exclusion Criteria:

1. A time interval between treatment and image examination greater than 1 month;
2. A history of other malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients with PET/CT or CT examination before any cancer-specific treatment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2012-2021
  The interval between the date of diagnosis and death

SECONDARY OUTCOMES:
Progression free survival | 2012-2021
  The interval between the date of treatment initiation and disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China